CLINICAL TRIAL: NCT03530189
Title: Neurodevelopmental Outcome of Very Preterm Infants With Glucose Level Disturbances at the Age of Two
Brief Title: Outcome of Very Preterm Infants With Glucose Level Disturbances
Status: Completed | Type: Observational
Sponsor: University Hospital Rijeka (Other)
Responsible Party: Principal Investigator, Ivona Butorac Ahel, Ivona Butorac Ahel, MD, MS, principal investigator, University Hospital Rijeka
Other Study IDs: istrazivanje01
Record Dates: First submitted 2018-04-22; First posted 2018-05-21 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Cerebral Palsy Infantile
Keywords: Hyperglycemia;; Hypoglycemia;; Neurodevelopment;; Prematurity
MeSH Terms: conditions — Cerebral Palsy; Hyperglycemia; Hypoglycemia; Premature Birth | interventions — Glucose; Insulin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normoglycemic group: The infant will enter this group if a single blood glucose concentration is between 2.1 and 2.5 mmol/l (38-45 mg/dL), or a single blood glucose concentration is between 8.6 - 10 mmol/l (155-180 mg/dL) with all other measures between 2.6 and 8.5 mmol/l (47-153 mg/dL).
  To all premature infants intravenous 10% dextrose at 60-90 mL/kg/day will be started as soon as possible after birth.
  Interventions: Drug: 10% dextrose
- Group with impaired glucose: The infant can be hypoglycemic, hyperglycemic or unstable. The infant will be hypoglycemic if blood glucose concentration is ≤2,5 mmol/l (45 mg/dL) on ≥2 measures >1 hour apart, or any blood glucose concentration is≤2,0 mmol/l (36 mg/dL). Hypoglycemia will be treated with intravenous bolus of 10% dextrose.
  The infant will be hyperglycemic if blood glucose concentration is ≥8,6 mmol/l (155 mg/dL) on ≥2 measures >1 hour apart, or any blood glucose concentration ≥10,1 mmol/l (182 mg/dL). Hyperglycemia will be managed by reducing the glucose infusion rate or initiation of an insulin infusion.
  The infant will be unstable if at least 1 blood glucose concentration is ≤2,5 mmol/l (45 mg/dL) and ≥1 blood glucose concentration is ≥8,6 mmol/l (155 mg/dL).
  Interventions: Drug: bolus of dextrose, reducing the glucose infusion, insulin

INTERVENTIONS:
Drug: 10% dextrose — After birth the intravenous 10% dextrose at 60-90 ml/kg/day will be started as soon as possible
  Other Names: There is no other intervention names
  Groups: Normoglycemic group
Drug: bolus of dextrose, reducing the glucose infusion, insulin — Hypoglycemia will be treated with 2 mL/kg to 3 mL/kg (200-300 mg/kg) intravenous bolus of 10% dextrose.
  Hyperglycemia will be managed by reducing the glucose infusion rate or initiation of an insulin infusion.
  Other Names: There is no other intervention names
  Groups: Group with impaired glucose

SUMMARY:
The hypothesis of this prospective, cohort study is that hyperglycemia, hypoglycemia and unstable glucose levels in the first seven days of life in infants born very preterm and at very low birth weights can harm long-term neurodevelopment. The objective of the study is to investigate the relationship between early neonatal glycemia, neonatal characteristics, and developmental outcomes in preterm infants. All infants born before 32. gestational week or below 1500 g admitted to the neonatal intensive care unit will be included in the study. According to the glucose values, the infants will be divided into the normoglycemic group and the group with disturbed glucose concentration. In the corrected age of two neurodevelopmental outcome will be assessed and categorized as normal, mild, moderate or severe impairment. Since the results of published studies about the effects of asymptomatic neonatal hypoglycemia and hyperglycemia on neurodevelopment are inconsistent, the correlation between early disturbances in glucose levels and neurodevelopmental outcome will be assessed.

DETAILED DESCRIPTION:
All infants born before 32 weeks of gestation or weighing <1500 g and admitted to the Neonatal intensive care unit of the University Hospital Center Rijeka will be included into the study. The investigators will collect data from the neonatal period, including: gestational age, sex, birth weight, Apgar score at 1 and 5 minutes, socioeconomic status and Clinical Risk Index for Babies scoring system (CRIB II). Blood glucose levels will be measured at 3rd, 12th, and 18th hour after birth on the first day of life, and from the 2nd to the 7th day of life blood glucose levels will be measured once a day. According to the blood glucose concentrations infants will be divided into normoglycemic group and group with disturbed glucose concentration. The relationship between glycemia category and 2-year outcomes will be investigated. In the corrected age of two years neurodevelopmental outcome will be assessed. Certified psychologists will assess cognitive, motor and language development with the Bayley Scales of Infant and Toddler Development (Bayley III). Bayley III scales are standardized to a mean (SD) score of 100. Pediatric neurologists or pediatrics will examine the children and will estimate the neuromotor function. Cognitive, motor and language development were considered normal if the composite score on the respective Bayley-III score was ≥mean -1SD; mildly impaired if the score was < -1 SD and ≥ -2 SD; moderately impaired if the score was <-2 SD and ≥3 SD; and severely impaired if the score was < mean -3SD.

Cerebral palsy (CP) was evaluated according to the European Cerebral Palsy Network definition. The severity of CP was classified as mild in children who were able to walk without an aid, moderate in children able to walk with an aid, and severe in children who were unable to walk even with an aid.

Children unable to fixate and follow a light with either eye were considered bilaterally blind. Children registered at low-vision centers without blindness were recorded as having moderate visual impairment. Severe auditory impairment was defined as hearing loss that could not be corrected with a hearing aid and moderate auditory impairment was defined as hearing loss corrected with a hearing aid.

The overall outcome was categorized as normal, mild, moderate or severe impairment. Mild impairment was defined as scores between -1and -2 standard deviations from the mean of any of the Bayley-III scales or mild CP. Moderate impairment was defined as scores between -2and -3 standard deviations from the mean of any of the Bayley-III scales, moderate CP, or moderate visual or hearing impairment. Severe impairment was defined as scores between < mean -3 standard deviations of any of the Bayley-III scales, severe CP, or bilateral blindness or deafness.

ELIGIBILITY:
Inclusion Criteria:

* infants born weighing <1500 g or at <32 weeks of gestation

Exclusion Criteria:

* infants with significant congenital abnormalities
* infants died before day 7
* infants whose mothers suffer from type 1, type 2 diabetes mellitus or gestational diabetes

Ages: 24 Weeks to 27 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: We will include all infants born before 32 of weeks gestation or weighing below 1500 g and admitted to the Neonatal intensive care unit (NICU) of University Hospital Center Rijeka. Blood glucose concentrations will be measured and recorded from birth until the end of postnatal day 7. Based on the values of glucose concentrations, infantsi will be categorized as normoglycemic, hypoglycemic, hyperglycemic and unstable. At the age between 22,5 and 26,5 months of corrected age assessment by neurologist and psychologist will be performed.
  This study is approved by Ethics Committee of University Hospital Center Rijeka and by the Ethics Committee of University of Rijeka - Faculty of Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Neurodevelopmental outcome of each group at the age of two performed using Bayley Scales of Infant and Toddler Development Bayley III | up to 27 months
  Mild impairment was defined as scores between -1and -2 standard deviations (70 - 85) from the mean of any of the Bayley-III scales or mild CP. Moderate impairment was defined as scores between -2and -3 standard deviations (55 - 70) from the mean of any of the Bayley-III scales, moderate CP, or moderate visual or hearing impairment. Severe impairment was defined as scores between < mean -3 standard deviations (<55) of any of the Bayley-III scales, severe CP, or bilateral blindness or deafness.

CONTACTS AND LOCATIONS:
Overall Officials: Ivona Butorac Ahel, MD, MS, Principal Investigator — University Hospital Center Rijeka, 51 000 Rijeka, Croatia
Locations (1):
- University Hospital Center Rijeka, Rijeka, Croatia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tottman AC, Alsweiler JM, Bloomfield FH, Gamble G, Jiang Y, Leung M, Poppe T, Thompson B, Wouldes TA, Harding JE; PIANO Study Group. Long-Term Outcomes of Hyperglycemic Preterm Infants Randomized to Tight Glycemic Control. J Pediatr. 2018 Feb;193:68-75.e1. doi: 10.1016/j.jpeds.2017.09.081. Epub 2017 Dec 1. PMID 29198539
- [Background] Sinclair JC, Bottino M, Cowett RM. Interventions for prevention of neonatal hyperglycemia in very low birth weight infants. Cochrane Database Syst Rev. 2011 Oct 5;(10):CD007615. doi: 10.1002/14651858.CD007615.pub3. PMID 21975772
- [Background] Mitanchez D. Glucose regulation in preterm newborn infants. Horm Res. 2007;68(6):265-71. doi: 10.1159/000104174. Epub 2007 Jun 20. PMID 17587854
- [Background] Goode RH, Rettiganti M, Li J, Lyle RE, Whiteside-Mansell L, Barrett KW, Casey PH. Developmental Outcomes of Preterm Infants With Neonatal Hypoglycemia. Pediatrics. 2016 Dec;138(6):e20161424. doi: 10.1542/peds.2016-1424. Epub 2016 Nov 4. PMID 27940690
- [Background] Tin W, Brunskill G, Kelly T, Fritz S. 15-year follow-up of recurrent "hypoglycemia" in preterm infants. Pediatrics. 2012 Dec;130(6):e1497-503. doi: 10.1542/peds.2012-0776. Epub 2012 Nov 5. PMID 23129080
- [Background] Lucas A, Morley R, Cole TJ. Adverse neurodevelopmental outcome of moderate neonatal hypoglycaemia. BMJ. 1988 Nov 19;297(6659):1304-8. doi: 10.1136/bmj.297.6659.1304. PMID 2462455
- [Background] Hey E. Hyperglycaemia and the very preterm baby. Semin Fetal Neonatal Med. 2005 Aug;10(4):377-87. doi: 10.1016/j.siny.2005.04.008. PMID 15927546
- [Background] Decaro MH, Vain NE. Hyperglycaemia in preterm neonates: what to know, what to do. Early Hum Dev. 2011 Mar;87 Suppl 1:S19-22. doi: 10.1016/j.earlhumdev.2011.01.005. Epub 2011 Jan 26. PMID 21276670
- [Background] Surveillance of Cerebral Palsy in Europe. Surveillance of cerebral palsy in Europe: a collaboration of cerebral palsy surveys and registers. Surveillance of Cerebral Palsy in Europe (SCPE). Dev Med Child Neurol. 2000 Dec;42(12):816-24. doi: 10.1017/s0012162200001511. PMID 11132255